CLINICAL TRIAL: NCT02217670
Title: Comparative Bioavailability Study of Metformin HCl 1000 mg Granules vs Glucophage 1000 mg Film-coated Tablet
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Commercial reasons
Sponsor: Disphar International B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: METF-GT016
Record Dates: First submitted 2014-08-14; First posted 2014-08-15 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2016-01

CONDITIONS: Comparative Bioavailability
MeSH Terms: interventions — Metformin

ARMS (2):
- Metformin (test) (Experimental): single oral dose of Metformin 1000 mg granules
  Interventions: Drug: Metformin 1000 mg granules
- Metformin (reference) (Active Comparator): Single dose of Glucophage 1000 mg film-coated tablet
  Interventions: Drug: Metformin 1000 mg film-coated tablets

INTERVENTIONS:
Drug: Metformin 1000 mg granules
  Arms: Metformin (test)
Drug: Metformin 1000 mg film-coated tablets
  Other Names: Glucophage
  Arms: Metformin (reference)

SUMMARY:
The main purpose of this study is to assess comparative bioavailability of a test formulation of Metformin HCl 1000 mg granules manufactured by Indeus Life Sciences Pvt. Ltd., Mumbai India (An Affiliate Of Disphar International B.V., The Netherlands) relative to Glucophage 1000 mg film-coated tablets of Merck GmbH, Austria in 54 healthy adult subjects under fed conditions. The second aim is to asses the safety of subjects and to determine other pharmacokinetic data.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 50 years, inclusive.
2. Body Mass Index (BMI) range is within 18.5 - 30.0 Kg/m2.
3. Subject does not have a known allergy to the drug under investigation or any of its ingredients or any other related drugs.

Exclusion Criteria:

1. Medical demographics performed not longer than two weeks before the initiation of the clinical study with significant deviations from the normal ranges.
2. Results of laboratory tests which are outside the normal range or HbA1c test or liver or kidney function tests (Creatinine levels and ALP will be accepted if below reference range) that are outside the reference range or Hb or RBC indices (MCV, MCH, MCHC) with deviation outside 5% of the reference range.
3. Acute infection within one week preceding first study drug administration.
4. History of drug or alcohol abuse.
5. Subject is a heavy smoker (more than 10 cigarettes per day).
6. Subject does not agree not to take any prescription or non-prescription drugs within the two weeks preceding the first study drug administration until donating the last sample of the study.
7. Subject does not agree not to take any vitamins taken for nutritional purposes within two days before first study drug administration until donating the last sample of the study.
8. Subject is on a special diet (for example subject is a vegetarian).
9. Subject consumes large quantities of alcohol or beverages containing methylxanthines e.g. caffeine (coffee, tea, cola, chocolate etc).
10. Subject does not agree not to consume any beverages or food containing alcohol 48 hours prior to study drug administration until donating the last sample in each respective period.
11. Subject does not agree not to consume any beverages or food containing methyl-xanthines e.g. caffeine (coffee, tea, cola, chocolate etc.) 24 hours prior to the study drug administration until the end of confinement period.
12. Subject does not agree not to consume any beverages or food containing grapefruit 7 days prior to first study drug administration until donating the last sample in the study.
13. Subject has a history of severe diseases which have direct impact on the study.
14. Participation in a bioequivalence/bioavailability study or in a clinical study within the last 80 days before first study drug administration.
15. Subject intends to be hospitalized within 3 months after first study drugs administration.
16. Subjects who donated blood or its derivatives in the past 3 months or who through completion of this study, would have donated more than 1250 ml in 120 days, 1500 ml in 180 days, 2000 ml in 270 days, 2500 ml of blood in 1 year.
17. The female subject is pregnant or lactating.
18. Subject has a history of significant asthma, peptic or gastric ulcer, sinusitis, pharyngitis, renal disorder (impaired renal function), hepatic disorder (impaired hepatic function), cardiovascular disorder, neurological disease such as epilepsy, haematological disorders, type I diabetes or diabetic ketoacidosis, lactic acidiosis, Vitamin B12 deficiency, psychiatric, dermatologic, immunological disorders or surgery.
19. Subject does not agree not to engage in strenuous exercise at least one day prior to study drug administration.
20. Subject having at screening examination a pulse outside the normal range of (60-100 beat per minute) or a body temperature outside the normal range of (36.4-37.7 ○C) or a respiratory rate outside the normal range of (14-20 breath per minute) or a sitting blood pressure less than 100/60 mm Hg or more than or equal to 140/90 mm Hg.
21. Subject has history of difficulties in swallowing or any gastrointestinal disease which could affect the drug absorption.
22. Subject undergoing radiologic studies involving intravascular administration of iodinated contrast materials (for example, intravenous urogram, intravenous cholangiography, angiography, and computed tomography (CT) scans with intravascular contrast materials).
23. Fasting blood sugar at screening is less than 70 mg/dl.
24. Subject has diabetes mellitus.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
AUC(0-t) | Before dosing (0.00 hour) and at the following times after the dose: 0.33, 0.66, 1.00, 1.33, 1.66, 2.00, 2.33, 2.66, 3.00, 3.33, 3.66, 4.00, 5.00, 6.00, 8.00, 12.00, 16.00 and 24.00 hours.
Cmax | Before dosing (0.00 hour) and at the following times after the dose: 0.33, 0.66, 1.00, 1.33, 1.66, 2.00, 2.33, 2.66, 3.00, 3.33, 3.66, 4.00, 5.00, 6.00, 8.00, 12.00, 16.00 and 24.00 hours.

SECONDARY OUTCOMES:
tmax | Before dosing (0.00 hour) and at the following times after the dose: 0.33, 0.66, 1.00, 1.33, 1.66, 2.00, 2.33, 2.66, 3.00, 3.33, 3.66, 4.00, 5.00, 6.00, 8.00, 12.00, 16.00 and 24.00 hours.
AUC(0-inf) | Before dosing (0.00 hour) and at the following times after the dose: 0.33, 0.66, 1.00, 1.33, 1.66, 2.00, 2.33, 2.66, 3.00, 3.33, 3.66, 4.00, 5.00, 6.00, 8.00, 12.00, 16.00 and 24.00 hours.
AUCres | Before dosing (0.00 hour) and at the following times after the dose: 0.33, 0.66, 1.00, 1.33, 1.66, 2.00, 2.33, 2.66, 3.00, 3.33, 3.66, 4.00, 5.00, 6.00, 8.00, 12.00, 16.00 and 24.00 hours.
t1/2 | Before dosing (0.00 hour) and at the following times after the dose: 0.33, 0.66, 1.00, 1.33, 1.66, 2.00, 2.33, 2.66, 3.00, 3.33, 3.66, 4.00, 5.00, 6.00, 8.00, 12.00, 16.00 and 24.00 hours.

OTHER OUTCOMES:
Number of participants with adverse events. | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- International Pharmaceutical Research Center, Amman, Jordan